CLINICAL TRIAL: NCT02620501
Title: Does Topical Lidocaine Reduce The Amount of Intravenous Conscious Sedation Required To Complete Diagnostic Upper Endoscopy and Shorten Recovery Time? A Double Blinded, Randomized, Placebo Controlled Study.
Brief Title: Does Use of Topical Lidocaine in EGD Reduce Amount of IV Midazolam and Fentanyl Required and Shorten Recovery Time
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Adam Tritsch, Gastroenterology Fellow, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BrookeAMC
Record Dates: First submitted 2015-01-26; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Dysphagia; GERD; Abdominal Pain
Keywords: EGD; topical lidocaine; recovery time; intravenous sedation
MeSH Terms: conditions — Deglutition Disorders; Gastroesophageal Reflux; Abdominal Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Patients will receive 10cc of 1/2 normal saline to gargle prior to EGD
  Interventions: Drug: Placebo
- Experimental (Experimental): Patients will receive 10cc of 2% topical lidocaine to gargle prior to EGD
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — topical lidocaine
  Arms: Experimental
Drug: Placebo — 0.45% Normal Saline
  Arms: Placebo

SUMMARY:
Patients will be randomized to a placebo or study group who will receive topical lidocaine prior to EGD. Amount of medication used, recovery time, patient/endoscopist satisfaction will then be assessed.

DETAILED DESCRIPTION:
The study will be a double blinded randomized placebo controlled trial

Patients between 18 and 89 years old who are scheduled for EGD may be eligible to enroll in the study. Potential subjects will be sought through referral by their treating attending and fellow gastroenterologist, who will be apprised of the inclusion and exclusion criteria. Patients possibly meeting inclusive and exclusive criteria will be approached and discussed the study further with the investigators. Those expressing a desire to participate in the study will be given written informed consent prior to participation. The investigators will enroll patients into the study with a goal of at least 53 patients in each group which is the number of patients our statistician recommended to appropriately power our study.

Patients who consent to enroll in the study will be randomized into 2 groups. Group 1: Swish and swallow 10ml of 2% lidocaine solution Group 2: Swish and swallow 10ml of 0.45% sodium chloride solution

The patients will then undergo endoscopy for the indication identified in their clinic appointment. Following the procedure, patients will be taken to the recovery area and recovered per clinic protocol. The endoscopist will complete a satisfaction questionnaire. The day following the procedure a nurse will call to check for post-operative complications per clinic protocol. The day following, an investigator will also call to perform a patient satisfaction survey..

ELIGIBILITY:
Inclusion Criteria:

* EGD alone performed by staff gastroenterologist as an outpatient
* Between the age of 18 and 89
* Not requiring anesthesia support or use of medications other than fentanyl and midazolam

Exclusion Criteria:

* Prior history of head and neck surgery
* Known hypersensitivity to local anesthetics, the amide type or any components of the topical lidocaine
* Patients having interventions other than polypectomy performed
* Pregnant or breast feeding females
* Patients with severe liver impairment
* Known hypersensitivity to benzodiazepine or fentanyl

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-02 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Amount of sedation used | 60 minutes
  We will record the amount of sedation used during the procedure

SECONDARY OUTCOMES:
Recovery time | 120 minutes
  We will record the amount of time it takes to recover following the procedure
Patient and physician satisfaction | 24 hours
  We will assess patient and physician satisfaction with the procedure through use of a questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Adam M Tritsch, MD, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

REFERENCES:
- [Background] Davis DE, Jones MP, Kubik CM. Topical pharyngeal anesthesia does not improve upper gastrointestinal endoscopy in conscious sedated patients. Am J Gastroenterol. 1999 Jul;94(7):1853-6. doi: 10.1111/j.1572-0241.1999.01217.x. PMID 10406247